CLINICAL TRIAL: NCT06093321
Title: A Randomized, Blinded, Active-Controlled, Matched Pairs, Single-Institution, Non-Inferiority Trial to Compare and Evaluate the Efficacy and Safety of SYB PDO Thread and MINT Lift® for Temporarily Improvement of Nasolabial Folds
Brief Title: A Study Comparing SYB PDO Thread and MINT Lift® for Temporary Nasolabial Fold Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR_PDO_301
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-10

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Intervention Model Description: A Randomized, Subject-Independent Rater blinding, Paired Matching, Active-Controlled, Single Institution, Non-Inferiority Pivotal Trials
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYB PDO Thread (Experimental): PDO Thread
  Interventions: Device: SYB PDO Thread
- MINT lift® (Active Comparator): PDO Thread
  Interventions: Device: MINT lift®

INTERVENTIONS:
Device: SYB PDO Thread — Apply the test device (SYB PDO Thread) and the control device (MINT lift®) with 7±1 lines on each side of the nasolabial fold.
  Arms: SYB PDO Thread
Device: MINT lift® — Apply the test device (SYB PDO Thread) and the control device (MINT lift®) with 7±1 lines on each side of the nasolabial fold.
  Arms: MINT lift®

SUMMARY:
The objective of this clinical trial is to verify the safety and efficacy of SYB PDO Thread in the temporary improvement of nasolabial Folds.

ELIGIBILITY:
Inclusion Criteria:

1. Those desiring temporary improvement of central facial nasolabial folds and having a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4.
2. Individuals willing to discontinue all dermatological procedures or treatments, including wrinkle improvement in the central facial nasolabial fold, throughout the duration of this clinical trial.

Exclusion Criteria:

1. Individuals who need to take anticoagulants from 2 weeks before the application of the clinical trial medical device to 2 weeks after (low-dose aspirin 100mg, maximum 300mg/day, is allowed).
2. Those who need to take Vitamin E supplements, NSAIDs, or collagen supplements from 1 week before the application of the clinical trial medical device to 1 week after.
3. Individuals with a history of bleeding disorders, either past or present.
4. Those who have received treatments such as deep chemical peels, skin rejuvenation procedures, plastic surgery (including Botox injections), wrinkle improvement, or acne scar treatment on the face within 24 weeks from the screening date.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants with a minimum 1-point improvement in WSRS scores, as evaluated by independent rater 3 months after device application. | 3months
  The Wrinkle Severity Rating Scale is a 5-point scale with 1 = Absent; 2 = Mild; 3 = Moderate; 4 = Severe and 5 = Extreme. 1 is the best outcome while 5 is the worst outcome. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Park, M.D.,Ph.D., Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea